CLINICAL TRIAL: NCT04058262
Title: Impact of Meditation and Reiki on Assisted Reproduction Techniques Outcomes: a Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Impact of Meditation and Reiki on Assisted Reproduction Techniques Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13851019.9.0000.5149
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Infertility
Keywords: in vitro fertilization; assisted reproduction; pregnancy rate; meditation; Reiki
MeSH Terms: conditions — Infertility | interventions — Therapeutic Touch; Meditation; Amyloid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meditation presential (Experimental)
  Interventions: Other: Meditation presential
- Reiki (Experimental)
  Interventions: Other: Reiki
- Meditation (app) (Experimental)
  Interventions: Other: Meditation (app)
- round of conversation (Placebo Comparator)
  Interventions: Other: round of conversation

INTERVENTIONS:
Other: Meditation presential — Facilitator-guided meditation in groups or individually, in 45-minute sessions twice a week for 2 weeks, in a quiet room with controlled light and temperature, and comfortable cushions and chairs.
  Arms: Meditation presential
Other: Reiki — Reiki will be performed in 45-minute sessions twice a week for 2 weeks then in a quiet room with controlled brightness and temperature.
  Arms: Reiki
Other: Meditation (app) — Mindfulness meditation guided through 10-15 minute audio using app, to be practiced daily at home.
  Arms: Meditation (app)
Other: round of conversation — The Round of Conversation will take place twice a week, lasting 45 minutes, for two weeks thereafter, at the same clinic, where women will talk about their lives, their needs, how they handle reported situations and how also your skills and preferences.
  Arms: round of conversation

SUMMARY:
Infertility is estimated to affect 15% of reproductive age couples worldwide and is defined as the inability to conceive after 12 months of unprotected sex for women under 35 or 6 months for women over 35 and is associated with stress, especially due to psychological factors such as anxiety, frustration and depression. In addition, women seeking treatment for pregnancy suffer additional stressors - significant emotional burdens and physical changes that can increase stress and anxiety levels. The possibility of an association between emotional stress and pregnancy outcome in women undergoing assisted reproduction treatment makes important therapies that address the psychological state of these women. Meditation and Reiki have been used to successfully reduce stress and anxiety in various health contexts.

Reiki is a complementary health approach in which practitioners lightly place their hands on or just above a person to facilitate their own healing response. Reiki has been used as an adjunctive therapy to treat the symptoms common to infertile women seeking treatment, including anxiety, stress, depression, anger, despair and depression. Reviews of randomized controlled trials concluded that implementation of the Reiki intervention in health centers resulted in mental health benefits, including reduced tension, mental confusion, anxiety and pain as well as improved quality of life.

Meditation can be defined as a form of mental training aimed at improving an individual's psychological capacities, such as attentional and emotional self-regulation. Meditation encompasses a family of practices that include mindfulness meditation, mantra meditation, yoga, tai chi and chi gong. Meditation has been used specifically in women undergoing IVF treatment to successfully reduce symptoms related to psychological distress. Studies measure the development of self-compassion, mechanisms of emotion regulation, and coping strategies related to infertility and quality of life in infertility. However, only one study showed a relationship between meditation and pregnancy rate. Unfortunately, the authors incorporated yoga and psychological approaches into meditation. Therefore, we designed this study to evaluate the impact of Meditation and Reiki on the outcome of assisted reproduction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women submitted to Embryo Transfer
* Signed informed consent form
* Fresh or Frozen Embryo Transfer

Exclusion Criteria:

* No agreement to participate
* no embryo transfer
* surrogate embryo transfer

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 12 weeks
  presence of a gestational sac at 12 weeks of pregnancy

SECONDARY OUTCOMES:
stress levels | 3 weeks
  Stress evaluation using questionnaires DASS-21 (Depression, Anxiety and Stress Score) and/or PGWB-1 (Psichological General Well-being Index)

CONTACTS AND LOCATIONS:
Locations (1):
- ORIGEN - Centre for Reproductive Medicine, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Long L, Liu Y, He W, Li M. Effects of a mindfulness-based intervention on fertility quality of life and pregnancy rates among women subjected to first in vitro fertilization treatment. Behav Res Ther. 2016 Feb;77:96-104. doi: 10.1016/j.brat.2015.12.010. Epub 2015 Dec 19. PMID 26742022
- [Result] Nery SF, Paiva SPC, Vieira EL, Barbosa AB, Sant'Anna EM, Casalechi M, Dela Cruz C, Teixeira AL, Reis FM. Mindfulness-based program for stress reduction in infertile women: Randomized controlled trial. Stress Health. 2019 Feb;35(1):49-58. doi: 10.1002/smi.2839. Epub 2018 Oct 16. PMID 30328241
- [Derived] Nunes GM, Paiva SPC, Geber S, Serra ASVA, Sampaio MAC, Tavares RLC. The impact of extremely brief meditation and brief mindfulness interventions on assisted reproductive technologies success rates: A randomised controlled trial. Explore (NY). 2024 Nov-Dec;20(6):103067. doi: 10.1016/j.explore.2024.103067. Epub 2024 Sep 29. PMID 39374555